CLINICAL TRIAL: NCT03116321
Title: A Single Center, Single Dose, Open Label, Laboratory Blind, Randomized, Three Period, Six Sequence, Crossover Study to Determine the Bioequivalence of Two Different Sources of Eslicarbazepine Acetate (800 mg) and to Assess the Dose Equivalence of Two Different Dose Strengths of Eslicarbazepine Acetate (200 and 800 mg) in Healthy Subjects
Brief Title: Bioequivalence of Two Different Sources of Eslicarbazepine Acetate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-131
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test 1 - TBM (Treatment A - 1 × 800 mg tablet) (Experimental): single oral dose of 800 mg (1 × 800 mg tablet) of Eslicarbazepine acetate (ESL) as tablets, on each of three separate occasions, under fasting conditions.
  Route of administration:Oral.
  Interventions: Drug: Eslicarbazepine acetate (ESL)
- Test 2 - TBM (Treatment B - 2 × 200 mg tablet) (Experimental): single oral dose of 800 mg (4 × 200 mg tablet) of Eslicarbazepine acetate (ESL) as tablets, on each of three separate occasions, under fasting conditions.
  Route of administration:Oral.
  Interventions: Drug: Eslicarbazepine acetate (ESL)
- Reference Product - MF (Treatment C - 1 × 800 mg tablet) (Active Comparator): single oral dose of 800 mg (1 × 800 mg tablet) of Eslicarbazepine acetate (ESL) as tablets, on each of three separate occasions, under fasting conditions.
  Route of administration:Oral.
  Interventions: Drug: Eslicarbazepine acetate (ESL)

INTERVENTIONS:
Drug: Eslicarbazepine acetate (ESL) — Oral Tablet of 800 mg and 200 mg of ESL
  Other Names: Zebinix®; Aptiom®; Exalief®; BIA 2-093

SUMMARY:
The purpose of this study is to determine whether the test product, eslicarbazepine acetate 800 mg tablets (test 1, To be marketed (TBM) Treatment A), and the reference product, eslicarbazepine acetate 800 mg tablets (current Active pharmaceutical ingredient (API) source - Marketed formulation (MF)) (Reference, Treatment C), are bioequivalent and to demonstrate dose equivalence between eslicarbazepine acetate 4 x 200 mg tablets (test 2, TBM Treatment B) and eslicarbazepine acetate 800 mg tablet (Reference).

DETAILED DESCRIPTION:
The study will comprise:

* Screening period of maximum 21 days before the first administration of the investigational medicinal product (IMP);
* Three treatment periods (each of which will include a profile period of 72 hours) separated by a wash out period of 7 calendar days (minimum number of days based on half-life of the analyte) to 14 calendar days (maximum number of days based on logistical arrangements) between consecutive administrations of the IMP, and
* A post study visit within 1 and 2 weeks of completion of the last treatment period of the study or within 72 hours of termination or withdrawal.

Subjects will be assigned randomly to treatment sequence according to randomization schedule, before the first administration of IMP.

Subjects will be admitted to the study center on Day -1 and will be allowed to leave 24 hours after dosing. Subjects have to return for the subsequent blood sample collections up to 72 hours after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 55 years of age (inclusive) at screening.
* Body mass index (BMI) between 18.5 and 30 kg/m2 (both inclusive).
* Body weight not less than 50 kg.
* Medical history, vital signs, physical examination, standard 12-lead electrocardiogram (ECG) and laboratory investigations must be clinically acceptable or within laboratory reference ranges for the relevant laboratory tests, unless the investigator considers the deviation to be irrelevant for the purpose of the study.
* Non smokers or mild to moderate smokers (≤ 10 cigarettes or pipes per day).
* Females, if:

  * Not of childbearing potential, e.g., has been surgically sterilized, undergone a hysterectomy, amenorrhea for ≥ 12 months and considered post-menopausal, Note: In postmenopausal women, the value of the serum pregnancy test may be slightly increased. This test will be repeated to confirm the results. If there is no increase indicative of pregnancy, the female will be included in the study.

OR

• Of childbearing potential, the following conditions are to be met: Negative pregnancy test. If this test is positive, the subject will be excluded from the study. In the rare circumstance that a pregnancy is discovered after the subject received IMP, every attempt must be made to follow her to term.

Not lactating. Abstaining from sexual activity (if this is the usual lifestyle of the subject) or must agree to use an accepted method of contraception, and agree to continue with the same method throughout the study.

Examples of reliable methods of contraception include non hormonal intrauterine device and barrier methods combined with an additional contraceptive method.

In this study the concomitant use of hormonal contraceptives is NOT allowed. Other methods, if considered by the investigator as reliable, will be accepted (after discussion with sponsor medical monitor).

* Males must agree to use an accepted method of contraception with a pregnant partner or partner of childbearing potential (barrier methods combined with an additional contraceptive method, true abstinence or vasectomy) throughout the study and refrain from donating sperm throughout the study.
* Written consent given for participation in the study before any study-specific screening procedure is performed.

Exclusion Criteria:

* Evidence of psychiatric disorder, antagonistic personality, poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* Current alcohol use > 21 units of alcohol per week for males and > 14 units of alcohol per week for females. One unit (10 g alcohol) is equal to beer [330 mL], wine [200 mL], or distilled spirits [25 mL] per day.
* Regular exposure to substances of abuse or a history of alcoholism within 1 year prior to the first dose of IMP.
* Use of any medication, prescribed or over-the-counter or herbal remedies, within 2 weeks before the first administration of IMP except if this will not affect the outcome of the study in the opinion of the investigator. In this study the concomitant use of hormonal contraceptives is NOT allowed.
* Participation in another study with an experimental drug, where the last administration of the previous IMP was within 8 weeks (or within 5 elimination half-lives for chemical entities or 2 elimination half-lives for antibodies or insulin), whichever is the longer, before administration of IMP in this study, at the discretion of the investigator.
* Treatment within the previous 3 months before the first administration of IMP with any drug with a well-defined potential for adversely affecting a major organ or system.
* A major illness during the 3 months before commencement of the screening period.
* History of relevant hypersensitivity or allergy to any drug (including known hypersensitivity to the IMP, its excipients or to other carboxamide derivatives (e.g., carbamazepine, oxcarbazepine).
* History of bronchial asthma or any other bronchospastic disease.
* History of convulsions.
* History of porphyria.
* Relevant history or laboratory or clinical findings indicative of acute or chronic disease, likely to influence study outcome. The IMP is contraindicated in second or third degree atrioventricular block.
* Donation or loss of blood equal to or exceeding 500 mL during the 8 weeks before the first administration of IMP or received any blood or blood products.
* Diagnosis of hypotension made during the screening period. Supine systolic blood pressure should be at least 90/140 mmHg and diastolic BP 50/90 mmHg.
* Diagnosis of hypertension made during the screening period or current uncontrolled of hypertension.
* Resting pulse of > 100 beats per minute or < 40 beats per minute during the screening period, either supine or standing.
* Positive testing for human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C.
* Positive urine screen for drugs of abuse. In case of a positive result the urine screen for drugs of abuse may be repeated once at the discretion of the investigator.
* Positive pregnancy test.
* Males or females who plan to procreate during the study, or not willing to practice reliable forms of male or female contraception during the study and males who refuse to refrain from donating sperm throughout the study.
* Clinically relevant abnormalities in the coagulation tests.
* Clinically diagnosed peptic ulceration within the past 5 years.
* History of bleeding disorders.
* Vegetarian or any abnormal diet (for whatever reason).
* Difficulty in swallowing.
* Immunization using a live organism vaccine within 4 weeks before the first dosing of IMP.
* Any specific investigational product safety concern.
* Vulnerable subjects, e.g., persons in detention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-12-03 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | pre dose (0 hours) and at 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours post dose
  Primary Pharmacokinetic Parameters
Area under the plasma concentration versus time curve from time zero to t, where t is the time of the last quantifiable concentration (AUC(0-t)) | pre dose (0 hours) and at 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours post dose
  Primary Pharmacokinetic Parameters
Area under the plasma concentration versus time curve with extrapolation to infinity (AUC(0-t)) | pre dose (0 hours) and at 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours post dose
  Primary Pharmacokinetic Parameters

SECONDARY OUTCOMES:
Time to reach maximum observed plasma concentration (tmax) | pre dose (0 hours) and at 30 minutes, 1 hour, 1 hour 30 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours post dose
  Secondary Pharmacokinetic Parameters

IPD SHARING:
Plan to Share IPD: Undecided